CLINICAL TRIAL: NCT06551779
Title: Efficacy of Perineural Injection With Dextrose Versus Therapy Conventional Physics in Patients With Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celia Itxelt Infante Castro (Other Government)
Collaborators: ARIANA GUADALUPE MARTINEZ SILVA (Unknown); MARIA DE LOS ANGELES HERNANDEZ SANCHEZ (Unknown); MERCEDES DE JESUS JUAREZ LOPEZ (Unknown); IVAN HUERTA GRANADA (Unknown); MARIA CATALINA SANTIAGO SANTIAGO (Unknown); VICTOR MANUEL CAMARILLO NAVA (Unknown)
Responsible Party: Sponsor-Investigator, Celia Itxelt Infante Castro, Clinical Coordination of Health Education and Research., Instituto Mexicano del Seguro Social
Organization: Instituto Mexicano del Seguro Social (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-2024-1501-001
Record Dates: First submitted 2024-06-05; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Bell´s Palsy
Keywords: perineural injection therapy; dextrose; bell´s palsy; rehabilitation

STUDY DESIGN:
Intervention Model Description: Experimental Group: Patients who meet the inclusion and exclusion criteria, to whom perineural injection with dextrose and conventional physical therapy will be applied for the treatment of Bell's palsy.
  Control Group: Patients who meet the inclusion and exclusion criteria, to whom only conventional physical therapy will be applied for Bell's palsy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Baseline: Adequate assembly with balanced groups through randomization and clinical stratification.
  * Execution: Proper application of the experimental maneuver with established doses at each injection point.
  * Outcome: Same number of evaluations in both groups and a 20% increase in sample size in case of losses.
  * Masking: Triple-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grupo experimental: (Experimental): Experimental Group: Patients who meet the inclusion and exclusion criteria, to whom perineural injection with dextrose and conventional physical therapy will be applied for the treatment of Bell's palsy.
  Interventions: Procedure: inyección perineural con solución de dextrosa tamponada
- Control: (No Intervention): Control Group: Patients who meet the inclusion and exclusion criteria, to whom only conventional physical therapy will be applied for Bell's palsy.

INTERVENTIONS:
Procedure: inyección perineural con solución de dextrosa tamponada — Application of perineural injection with buffered dextrose solution, adding 2.5 ml of 7.5% sodium bicarbonate to a 250 ml bottle of glucose solution at 5% concentration, applying 1cc of the solution at different points on the path of the facial nerve.
  Arms: Grupo experimental:

SUMMARY:
Bell´s Palsy, a lower motor neuron injury that causes facial asymmetry due to facial weakness ranging from mild to total paralysis. Most of cases without determining a definitive established cause. The only authenticated findings are inflammation and edema of the facial nerve. In Mexico, it is among the first causes of medical attention. In the Mexican Clinical Practice Guide for Bells Palsy, thermotherapy, massage, and active exercises are recommended for its management. Perineural dextrose injection therapy (PIT) is a new treatment for peripheral neuropathy, which consists of injecting 5% buffered dextrose close to nerve pathways to restore nerve function and movement. Objective: Determine the effectiveness of perineural injection with dextrose versus conventional physical therapy for the treatment of patients with Bell´s palsy. Material and methods: Clinical trial, experimental, prolective, longitudinal, comparative and heterodemic. Resources and infrastructure: It will be carried out within the facilities of the Unidad de Medicina Física y Rehabilitación región centro. In human resources, doctors both specialists and residents in Rehabilitation Medicine and physical therapists. In material resources, stationery, for electroneuromyography study, perineural injection therapy, hand hygiene and disinfection, and for conventional rehabilitation therapy.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of dextrose perineural injection therapy while motivating and serving as a foundation for future studies to compare or create alternatives and therapeutic methods tailored to the needs patients, with the goal of improving functionality and aesthetics.

ELIGIBILITY:
* Inclusion Criteria: Patients with Bell's Palsy who:

  * Age 18 years and older.
  * Both male and female.
  * Duration of symptoms longer than 6 days.
  * Apparently healthy, without any associated comorbidities such as diabetes mellitus, obesity, hypothyroidism, hyperthyroidism, metabolic syndrome, or any neurological disorder.
  * Grade III (moderate dysfunction), IV (moderate to severe dysfunction), V (severe dysfunction), or VI (total paralysis) according to the House-Brackmann Classification.
  * Exclusive attention from UMF 2, 3, 4, 6, 11, 16, 29, 34, 35, 42, 94, 120 and the Physical Medicine and Rehabilitation Unit in the central region (employers and beneficiaries).
  * Exclusive attention from the UMF belonging to Mexico City (beneficiaries only).
  * Patients willing to participate in the study confirmed with signed informed consent.
* Exclusion Criteria:

  * Active smokers.
  * Patients with central facial paralysis.
  * Patients with peripheral facial paralysis secondary to tumors or surgical treatment.
  * Patients experiencing more than second episode of Peripheral Facial Paralysis.
  * Patients with cognitive and/or mental impairments.
  * Patients undergoing additional private therapy.
  * Patients with bilateral facial paralysis.
  * Pregnant patients.
  * Patients unwilling to participate in the study.
  * Patients who have received prior rehabilitation, laser, electrotherapy, or acupuncture.
* Elimination Criteria:

  * Patients who do not attend rehabilitation sessions.
  * Patients diagnosed with Sars-cov2 infection during the study.
  * Patients who discontinue treatment.
  * Patients developing other pathologies requiring special treatment.
  * Patients wishing to withdraw from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy in functionality | ≥8 weeks
  A= Functionality facial B= Recovery in time
Recovery in time | 1= ≥8 weeks 2= ≤ 8 weeks
  It is the action and effect of recovering or recovering (returning to oneself or to a normal state, take back what you had before, compensate) in a set time.
Functionality facial | ≥8 Weeks or ≤ 8 weeks
  1. Manual examination of facial muscles. It is a clinical evaluation to determine the function and strength of a person's facial muscles.
  2. Clinical evaluation. The House-Brackmann rating scale used to evaluate facial function and severity of facial paralysis peripheral, which consists of six levels to evaluate six facial expressions starting from normal (grade I) and as the last degree considers total paralysis (grade VI).
  3. Assessment electrophysiological with study of electroneurography of facial nerve that consists of the neuro conductions that they involve electrical stimulation of the nerve by measuring its motor response.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA DE LOS ANGELES HERNANDEZ SANCHEZ, DRA, Principal Investigator — MEDICA ADSCRITA A UNIDAD DE MEDICINA FISICA Y REHABILITACION REGION CENTRO IMSS
Locations (1):
- Unidad de Medicina Física Y Rehabilitacion Region Centro Imss, Mexico City, Cuauhtemoc, Mexico

IPD SHARING:
Plan to Share IPD: No